CLINICAL TRIAL: NCT00698256
Title: Effect of High Stanol Ester Dose on Serum Lipids, Carotenoids and Fat-soluble Vitamins
Acronym: maxsta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marjukka Kolehmainen (Other)
Collaborators: Raisio Plc (Industry)
Responsible Party: Sponsor-Investigator, Marjukka Kolehmainen, Senior scientist, University of Eastern Finland
Organization: University of Eastern Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 132\2007
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: vegetable oil-based spread and oat-based drink (no brand name available)
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: vegetable oil-based spread and oat-based drink (no brand name available)

INTERVENTIONS:
Dietary Supplement: vegetable oil-based spread and oat-based drink (no brand name available) — spread and drink (9 g stanols/d)
  Arms: 1
Dietary Supplement: vegetable oil-based spread and oat-based drink (no brand name available) — Spread and drink (not containing added stanols)
  Arms: 2

SUMMARY:
The aim was to investigate the effects of the consumption of high doses of plant stanol esters on concentrations of serum lipids, carotenoids and fat soluble vitamins. In addition, we investigated the metabolism of absorbed plant sterols from intestine without and with the consumption of plant stanol esters.

DETAILED DESCRIPTION:
Several studies have shown that 2-3 g of plant stanols as stanol esters reduce serum total and LDL cholesterol concentrations by 10-15%. There are only a few studies in which cholesterol-lowering effects of plant stanols have been studied with higher doses than that. In these studies with the stanol dose of 4 g/d no additional cholesterol-lowering effect has been reached. However, it would be interesting to know, how effective plant stanols are, if a dose is very high, or whether there is really a threshold effect in inhibition of cholesterol absorption. Plant sterols and stanols have been found to reduce serum β-carotene concentrations. Although they have not been shown to affect serum vitamin A concentrations, a concern has been aroused about safety of high doses of plant sterol and stanols. This is not unjustified, because the number of plant sterol and stanol containing products on the market continues to expand, and therefore, it is possible that the daily intake of plant sterols and stanols can rise very high.

In humans, the metabolism of plant sterols and stanols is not completely known. Recently, we showed that plant sterols are esterified in enterocytes as well as cholesterol facilitating their transport in lipoproteins. However, it is not known, how consumption of high doses of stanol esters affect the metabolism of plant sterols in enterocytes and their transport. This is important to know, when new foodstuffs enriched with plant sterols or stanols for cholesterol-lowering are developed.

In this study, the aim was to investigate the effects of the consumption of high doses of plant stanol esters on concentrations of serum lipids, carotenoids and fat soluble vitamins. In addition, we investigated the metabolism of absorbed plant sterols from intestine without and with the consumption of plant stanol esters.

Altogether 50 subjects with normo- or hypercholesterolemia (total cholesterol 4.5-7.5 mmol/l) were recruited to the study from an announcement in the local newspaper. The study is carried out with a randomized, double-blind and parallel design. The intervention group (n=25) consumes spread and oat drink enriched with plant stanol esters (9 g/d stanols) and the control group (n=25) the same product containing no added stanols for 10 weeks. The fasting blood samples are taken at weeks 0, 9, 10 and 14 (4 weeks after the end of the test product consumption). At week 10, an oral postprandial test is performed in 40 subjects in order to study the postprandial metabolism of plant sterols. From blood samples blood count and levels of serum liver enzymes (0 and 10 wk), concentrations of serum lipids, squalene and non-cholesterol sterols, α and β carotenoids, fat soluble vitamins A, E and D (0, 9 and 10 wk) and serum squalene and non-cholesterol sterols (14 wk) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol 4.5-7.5 mmol/l)
* Age 18-75 years

Exclusion Criteria:

* Liver, kidney and thyroid dysfunction
* Unstable coronary disease
* Inflammatory bowel disease
* Medication for hypercholesterolemia
* Plant stanol/sterol enriched foods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Serum lipids, Serum fat soluble vitamins and carotenoids, squalene and non-cholesterol sterols | baseline, at weeks 9, 10 and 14

CONTACTS AND LOCATIONS:
Locations (1):
- University of kuopio, Kuopio, Finland

REFERENCES:
- [Derived] Hallikainen M, Simonen P, Gylling H. Cholesterol metabolism and serum non-cholesterol sterols: summary of 13 plant stanol ester interventions. Lipids Health Dis. 2014 Apr 27;13:72. doi: 10.1186/1476-511X-13-72. PMID 24766766
- [Derived] Gylling H, Hallikainen M, Nissinen MJ, Miettinen TA. The effect of a very high daily plant stanol ester intake on serum lipids, carotenoids, and fat-soluble vitamins. Clin Nutr. 2010 Feb;29(1):112-8. doi: 10.1016/j.clnu.2009.08.005. Epub 2009 Aug 26. PMID 19709787